CLINICAL TRIAL: NCT02554617
Title: Measurements of Exhaled Nitric Oxide in Healthy Subjects in Thailand
Acronym: FeNO_nor
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Nualanong Visitsunthorn, Professor, Mahidol University
Other Study IDs: 555/2552(EC2)
Record Dates: First submitted 2010-07-18; First posted 2015-09-18 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Normal Non-fluency
Keywords: healthy people; fractional exhaled nitric oxide (FeNo); factors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine fractional exhaled nitric oxide (FeNO) level in healthy subjects among Thai populations.

DETAILED DESCRIPTION:
Fractional exhaled nitric oxide (FeNO) were produced from epithelial cells of inflammatory airways and eosinophils and this gas was discovered since 1991.

Fractional exhaled nitric oxide (FeNO) has direct association with severity of inflammation of bronchial trees and sputum eosinophils and use for additional investigation for diagnosis asthma or inflammatory airway diseases.

There are many factors from previous studies that associate with level of fractional exhaled nitric oxide (FeNO), one of that factors is race therefore we can't use level from another studies with different race for use as reference and there is no study about level of fractional exhaled nitric oxide in Thai population.

It is therefore desirable to examine level of fractional exhaled nitric oxide (FeNO) in healthy subjects among Thai population and will be the main objective of this research.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects in community

Exclusion Criteria:

* smoker or past history of smoking
* asthma, allergic rhinitis, chronic respiratory disease or other chronic illness
* history of wheezing within 12 months before enrollment
* history of upper or lower respiratory tract infection within 6 weeks before enrollment
* drink ethanol within 48 hours before enrollment
* drink caffeine within day before enrollment
* during pregnancy
* chronic use of any drugs
* participate other project within 30 days

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-10; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
fractional exhaled nitric oxide level | 10 minutes (average time ), on the day of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Professor Nualanong Visitsunthorn, MD, Principal Investigator — Department of Pediatrics, Faculty of Medicine Siriraj Hospital, Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok, Thailand